CLINICAL TRIAL: NCT00998127
Title: Patterns of Non-Adherence to Dual Anti-Platelet Regimen In Stented Patients: An Observational Single-Arm Study (The PARIS Registry)
Brief Title: Patterns of Non-Adherence to Dual Anti-Platelet Regimen In Stented Patients
Acronym: PARIS
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: GCO 10-1196; 09-367; 09-0421-F2L; 717/DG; AAAE0348
Record Dates: First submitted 2009-10-16; First posted 2009-10-20 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Medication Non-adherence; Stent Thrombosis
Keywords: Dual Anti-Platelet Therapy; Non-adherence; MACE; NACE
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this observational research study is to determine when and why patients discontinue, interrupt, or disrupt the regimen of anti-platelet medications prescribed following stent implantation, and to examine the relationship between specific patterns of non-adherence and patient outcomes.

DETAILED DESCRIPTION:
Anti-platelet medicines are the cornerstone of therapy in patients who present with acute coronary syndromes, including unstable angina, non-ST elevation myocardial infarction (NSTEMI), and ST elevation myocardial infarction (STEMI). Multiple clinical trials have demonstrated the efficacy of dual anti-platelet therapy (DAPT) for the prevention of thrombotic events in patients who present with unstable coronary symptoms; in particular, patients who are to receive percutaneous coronary intervention (PCI). Dual anti-platelet therapy consists of a combination of aspirin and a thienopyridine (such as clopidogrel or ticlopidine). While premature discontinuation (within the first 6 months) of such therapy is associated with an increased risk of stent thrombosis, the optimal duration of DAPT has not yet been precisely determined.

Although studies suggest an increased risk of stent thrombosis and adverse events within days after thienopyridine discontinuation, no study has collected detailed data as to the exact dates and reasons that anti-platelet agents were discontinued - thus, the true risks of premature early or even scheduled late discontinuation are unknown.

Furthermore, there are multiple modes that impact subject adherence to DAPT. These include non-compliance and cost issues.

We have determined three modes why subjects may not adhere to DAPT. These include:

* Discontinuation - These subjects have discontinued the use of DAPT (aspirin or thienopyridines) as per recommendation of their physician who has felt that the subject no longer needs this therapy.
* Interruption - These subjects have interrupted their DAPT use on a voluntary basis and under the guidance and recommendation of their physician due to the need for a surgical procedure, and will reinstitute the use of DAPT within 14 days of stopping the therapy. Interruptions must be guided by the physician/cardiologist taking care of the subject and not by other health care professionals.
* Disruption - These subjects have disrupted their DAPT use, either because of a bleeding episode (minor or major) or non-compliance. Non-compliance will include continued use of DAPT at lower dose levels than prescribed either through smaller daily doses or less frequent than daily use.

These modes have not previously been systematically collected and correlated with adverse clinical events such as stent thrombosis. Furthermore, the relation of events to subsequent disruption of DAPT has not been studied prospectively. Subjects enrolled in this registry will be followed for approximately 24 months to determine the incidence of adherence according to the above classification. All patients will have their events and DAPT use monitored during the follow-up period. The assumption is that most subjects will discontinue their therapy voluntarily (usually according to their physician's advice) and that it is only those with disrupted therapy who are at risk for major adverse cardiac events (MACE). This registry will examine the predictors of DAPT disruption based on subject's demographics and determine the relationship of bleeding versus MI in these subjects using a time-dependent covariate adjusted analysis. Finally, since there are two completely different categories within the disrupted group, (non-compliance vs. event driven disruption), we will examine these patients separately as well, as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* The subject has been informed of the nature of the study, agrees to its provisions, and has signed and been provided an "Informed Consent Form" approved by the appropriate Medical Ethics Committee (MEC) or Institutional Review Board (IRB).
* The subject must be ≥18 of age (or minimum age as required by local regulations) at the time of enrollment with successful stent placement in one or more lesions in native coronary arteries using an approved coronary stent.
* Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV), OR unstable angina pectoris (Braunwald Classification B&C, I-II-III), OR subjects with documented silent ischemia, OR acute myocardial infarction.
* The subject is willing and able to cooperate with the study procedures and required follow-ups.

Exclusion Criteria:

* Subjects with hypersensitivity or allergies to anti-platelet therapy.
* Subjects in whom anti-platelet and/or anticoagulation therapy is contraindicated.
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following the index procedure.
* The subject is participating in an investigational device or drug study. Subject must have completed the follow-up phase of any previous study at least 30 days prior to enrollment in this study.
* Subject has a history of bleeding diathesis or coagulopathy.
* Subject has other medical illness (e.g., cancer, known malignancy or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause non-compliance with the followups as defined by the protocol or confound the data interpretation.
* Evidence of stent thrombosis by visual angiographic assessment during the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects in any of the participating US or European sites who have undergone successful stent implantation in a native coronary artery.
Sampling Method: Non-Probability Sample
Enrollment: 5031 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Anti-platelet agent discontinuation/ interruption/ disruption | at 1 month
Incidence of Anti-platelet agent discontinuation/ interruption/ disruption | at 6 months
Incidence of Anti-platelet agent discontinuation/ interruption/ disruption | at 12 months
Incidence of Anti-platelet agent discontinuation/ interruption/ disruption | at 24 months
Incidence of major and minor bleeding (according to TIMI and ACUITY definitions) | at 1 month
Incidence of major and minor bleeding (according to TIMI and ACUITY definitions) | at 6 months
Incidence of major and minor bleeding (according to TIMI and ACUITY definitions) | at 12 months
Incidence of major and minor bleeding (according to TIMI and ACUITY definitions) | at 24 months
Incidence of definite and/or probable stent thrombosis (ARC definition) | at 1 month
Incidence of definite and/or probable stent thrombosis (ARC definition) | at 6 months
Incidence of definite and/or probable stent thrombosis (ARC definition) | at 12 months
Incidence of definite and/or probable stent thrombosis (ARC definition) | at 24 months

SECONDARY OUTCOMES:
Incidence of MACE. (MACE is defined as the composite of cardiac death, Q-wave myocardial infarction (MI), and unscheduled, ischemia driven revascularization of the target lesion.) | at 1 month
Incidence of MACE. (MACE is defined as the composite of cardiac death, Q-wave myocardial infarction (MI), and unscheduled, ischemia driven revascularization of the target lesion.) | at 6 months
Incidence of MACE. (MACE is defined as the composite of cardiac death, Q-wave myocardial infarction (MI), and unscheduled, ischemia driven revascularization of the target lesion.) | at 12 months
Incidence of MACE. (MACE is defined as the composite of cardiac death, Q-wave myocardial infarction (MI), and unscheduled, ischemia driven revascularization of the target lesion.) | at 24 months
Incidence of NACE (NACE is defined as the composite of cardiac death, MI (Q and non-Q-wave), ischemia driven revascularization of the target lesion and major bleeding (ACUITY criteria).) | at 1 month
Incidence of NACE (NACE is defined as the composite of cardiac death, MI (Q and non-Q-wave), ischemia driven revascularization of the target lesion and major bleeding (ACUITY criteria).) | at 6 months
Incidence of NACE (NACE is defined as the composite of cardiac death, MI (Q and non-Q-wave), ischemia driven revascularization of the target lesion and major bleeding (ACUITY criteria).) | at 12 months
Incidence of NACE (NACE is defined as the composite of cardiac death, MI (Q and non-Q-wave), ischemia driven revascularization of the target lesion and major bleeding (ACUITY criteria).) | at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Roxana Mehran, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Antonio Colombo, MD, Principal Investigator — San Raffaele Hospital (Milan, Italy)
Locations (15):
- United States (10):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Heart Center of Indiana, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Saint Luke's/ Mid-America Heart Institute, Kansas City, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Geisinger Medical Center Clinic, Danville, Pennsylvania
- Hopital Bichat, Paris, France
- Charite - Campus Benjamin Franklin, Berlin, Germany
- Onassis Cardiac Surgery Center, Athens, Greece
- Italy (2):
  - Careggi Hospital, Florence
  - San Raffaele Hospital, Milan

REFERENCES:
- [Derived] Baber U, Leisman DE, Cohen DJ, Gibson CM, Henry TD, Dangas G, Moliterno D, Kini A, Krucoff M, Colombo A, Chieffo A, Sartori S, Witzenbichler B, Steg PG, Pocock SJ, Mehran R. Tailoring Antiplatelet Therapy Intensity to Ischemic and Bleeding Risk. Circ Cardiovasc Qual Outcomes. 2019 Jan;12(1):e004945. doi: 10.1161/CIRCOUTCOMES.118.004945. PMID 30606052
- [Derived] Shah B, Baber U, Pocock SJ, Krucoff MW, Ariti C, Gibson CM, Steg PG, Weisz G, Witzenbichler B, Henry TD, Kini AS, Stuckey T, Cohen DJ, Iakovou I, Dangas G, Aquino MB, Sartori S, Chieffo A, Moliterno DJ, Colombo A, Mehran R. White Blood Cell Count and Major Adverse Cardiovascular Events After Percutaneous Coronary Intervention in the Contemporary Era: Insights From the PARIS Study (Patterns of Non-Adherence to Anti-Platelet Regimens in Stented Patients Registry). Circ Cardiovasc Interv. 2017 Sep;10(9):e004981. doi: 10.1161/CIRCINTERVENTIONS.117.004981. PMID 28916600
- [Derived] Baber U, Mehran R, Giustino G, Cohen DJ, Henry TD, Sartori S, Ariti C, Litherland C, Dangas G, Gibson CM, Krucoff MW, Moliterno DJ, Kirtane AJ, Stone GW, Colombo A, Chieffo A, Kini AS, Witzenbichler B, Weisz G, Steg PG, Pocock S. Coronary Thrombosis and Major Bleeding After PCI With Drug-Eluting Stents: Risk Scores From PARIS. J Am Coll Cardiol. 2016 May 17;67(19):2224-2234. doi: 10.1016/j.jacc.2016.02.064. Epub 2016 Apr 11. PMID 27079334
- [Derived] Mehran R, Baber U, Steg PG, Ariti C, Weisz G, Witzenbichler B, Henry TD, Kini AS, Stuckey T, Cohen DJ, Berger PB, Iakovou I, Dangas G, Waksman R, Antoniucci D, Sartori S, Krucoff MW, Hermiller JB, Shawl F, Gibson CM, Chieffo A, Alu M, Moliterno DJ, Colombo A, Pocock S. Cessation of dual antiplatelet treatment and cardiac events after percutaneous coronary intervention (PARIS): 2 year results from a prospective observational study. Lancet. 2013 Nov 23;382(9906):1714-22. doi: 10.1016/S0140-6736(13)61720-1. Epub 2013 Sep 1. PMID 24004642